CLINICAL TRIAL: NCT06284941
Title: A Study of Ropivacaine Complex Methylene Blue Fascia Iliaca Compartment Block on Analgesia in Patients Undergoing Hip Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wang wanxia (Other)
Responsible Party: Sponsor-Investigator, Wang wanxia, Principal Investigator, Yangzhou University
Organization: Yangzhou University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: KY 2023-001-001
Record Dates: First submitted 2024-02-04; First posted 2024-02-29 (Actual); Results first posted 2025-02-04 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-02

CONDITIONS: Femoral Neck Disease
MeSH Terms: interventions — Methylene Blue

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 0.25% ropivacaine 30ml for iliac fascia block (No Intervention)
- 0.25% ropivacaine+0.05% methylene blue 30ml for iliac fascia block (Experimental)
  Interventions: Drug: Ropivacaine combined with methylene blue for iliac fascia block

INTERVENTIONS:
Drug: Ropivacaine combined with methylene blue for iliac fascia block — Ultrasound guided iliac fascia block, administered with 30ml of 0.25% ropivacaine+0.05% methylene blue
  Arms: 0.25% ropivacaine+0.05% methylene blue 30ml for iliac fascia block

SUMMARY:
Total hip arthroplasty is currently the most effective method for treating hip joint lesions and improving quality of life, but postoperative severe pain is not conducive to rapid recovery of patients. In recent years, the widespread application of ultrasound has achieved good clinical results in iliac fascia block for postoperative analgesia in THA. However, the use of high-dose local anesthetics can increase the risk of local anesthetic poisoning, and the single block analgesia time is generally less than 24 hours. Methylene blue, as a long-acting analgesic drug, can block the pain transmission of nerve fibers for a long time, achieving analgesic effects without damaging neurons. This study used ultrasound-guided ropivacaine combined with methylene blue to perform iliac fascia block on patients undergoing total hip replacement, with the aim of prolonging pain relief time, reducing complications, and promoting postoperative recovery on the basis of traditional methods.

ELIGIBILITY:
Inclusion Criteria:

* Hip replacement surgery is indicated
* ASA Class II - Class III
* No history of analgesic or local anesthetic allergy
* No history of alcohol abuse or narcotic drug abuse
* Patients and their families have given informed consent and signed the informed consent form

Exclusion Criteria:

* Patient or family refusal to participate in the study
* Severe coagulation abnormalities
* Local anesthetic allergy
* Severe psychiatric illness or other communication disorder
* There is an infection at the puncture site
* History of neurological disease such as Guillain-Barré syndrome
* Delay in awakening post-surgery for more than 60 min,
* Post-surgical use of an analgesic pump
* Inability to follow-up at the required time points.

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 90 (Actual)
Dates: Start 2023-06-20 (Actual); Primary Completion 2024-02-28 (Actual); Study Completion 2024-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Zhang yang, Study Chair — not have
Locations (1):
- Jiangyan District Hospital of traditional Chinese medicine attached to the Nanjing University of Chinese Medicine, Taizhou, Jiangsu, China

REFERENCES:
- [Derived] Zhang Y, Yang S, Lu ZR, Zhou F, Liu MY. Analgesic effect of ropivacaine combined with methylene blue in fascia Iliaca block for patients undergoing hip arthroplasty. BMC Musculoskelet Disord. 2025 Mar 14;26(1):256. doi: 10.1186/s12891-025-08490-6. PMID 40087701

RESULTS

PARTICIPANT FLOW:
Groups:
- 0.25% Ropivacaine 30ml for Iliac Fascia Block: 0.25% ropivacaine 30ml for iliac fascia block
Period: Overall Study
Arm/Group | 0.25% Ropivacaine 30ml for Iliac Fascia Block | 0.25% Ropivacaine+0.05% Methylene Blue 30ml for Iliac Fascia Block
Started | 45 | 45
Completed | 45 | 45
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- 0.25% Ropivacaine 30ml for Iliac Fascia Block: Fascia iliaca block with ropivacaine: ultrasound-guided fascia iliaca block, administered with 30ml of 0.25% ropivacaine
- Total: Total of all reporting groups
Arm/Group | 0.25% Ropivacaine 30ml for Iliac Fascia Block | 0.25% Ropivacaine+0.05% Methylene Blue 30ml for Iliac Fascia Block | Total
Number analyzed (Participants) | 45 | 45 | 90
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 45 | 45 | 90
Age, Continuous [Mean (Standard Deviation); unit: Jiangyan District Hospital of traditiona] | 75.47 (5.54) | 73.93 (5.61) | 74.7 (5.60)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 32 | 62
  Male | 15 | 13 | 28
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 45 | 45 | 90
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  China | 45 | 45 | 90

OUTCOME MEASURES:

1. Primary Outcome: Visual Analogue Scale（VAS）
Description: Use a swimming ruler about 10 cm long, marked with 10 ticks on one side, and "0" and "10" at each end. A score of 0 indicates no pain, a score of 10 indicates the most severe pain that is unbearable, and the higher the score, the greater the degree of pain
Time Frame: From enrollment to 48 hours after surgery， the VAS scores at both rest and with activity (passive straight leg raise at 45°) were recorded at the following time points: before block and at 2, 6, 12, 24, and 48 h postoperatively
Measure: Median (Inter-Quartile Range); unit: score
Arm/Group | 0.25% Ropivacaine 30ml for Iliac Fascia Block | 0.25% Ropivacaine+0.05% Methylene Blue 30ml for Iliac Fascia Block
Number analyzed (Participants) | 45 | 45
score | 3.0 [2.0 to 3.5] | 4.0 [4.0 to 5.0]

2. Secondary Outcome: Hypersensitive C-reactive Protein
Description: Hypersensitive C-reactive protein, like procalcitonin, is an inflammatory marker. Both have the same meaning and are used to reflect the postoperative analgesic effect
Time Frame: From enrollment to 48 hours after surgery
Reporting Status: Not Posted

3. Secondary Outcome: Procalcitonin
Description: Procalcitonin is an inflammatory marker, which is associated with postoperative pain, the higher the degree of pain, the higher the procalcitonin value, the lower the pain level, and the lower the procalcitonin value, and the level of procalcitonin is used to reflect the postoperative analgesic effect
Time Frame: From enrollment to 48 hours after surgery
Reporting Status: Not Posted

4. Secondary Outcome: Neutrophil Lymphocyte Ratio
Time Frame: From enrollment to 48 hours after surgery
Reporting Status: Not Posted

5. Secondary Outcome: Mean Arterial Pressure
Time Frame: From entering the operating room to leaving the resuscitation room
Reporting Status: Not Posted

6. Secondary Outcome: Heart Rate
Time Frame: From entering the operating room to leaving the resuscitation room
Reporting Status: Not Posted

7. Secondary Outcome: Duration of Surgery
Time Frame: Intraoperative
Reporting Status: Not Posted

8. Secondary Outcome: Number of Postoperative Salvage Analgesia
Time Frame: From the end of surgery to 48 hours after surgery
Reporting Status: Not Posted

9. Secondary Outcome: Walking Distance for the First Time Getting Out of Bed
Time Frame: From the end of surgery to 48 hours after surgery
Reporting Status: Not Posted

10. Secondary Outcome: The Number of Activities of Getting Out of Bed 48 Hours After Surgery
Time Frame: From the end of surgery to 48 hours after surgery
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: The total time for collecting adverse events was approximately 48 hours, each participant was collected from the end of the surgery to 48h postoperatively.
Arm/Group | 0.25% Ropivacaine 30ml for Iliac Fascia Block | 0.25% Ropivacaine+0.05% Methylene Blue 30ml for Iliac Fascia Block
All-Cause Mortality (participants affected / at risk) | 0/45 | 0/45
Serious Adverse Events (participants affected / at risk) | 0/45 | 0/45
Other Adverse Events (participants affected / at risk) | 7/45 | 6/45
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 0.25% Ropivacaine 30ml for Iliac Fascia Block (N=45) | 0.25% Ropivacaine+0.05% Methylene Blue 30ml for Iliac Fascia Block (N=45)
Nausea and vomiting (Gastrointestinal disorders) | 7 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-12-24): https://cdn.clinicaltrials.gov/large-docs/41/NCT06284941/Prot_SAP_000.pdf